CLINICAL TRIAL: NCT00692016
Title: An Open Label, Randomized, Two-Way Crossover Study to Determine the Bioavailability of a Single, Oral Dose of an Extended Release Naproxen Sodium Tablet Under Fasting and Fed Conditions
Brief Title: Fast & Fed Pharmacokinetic (PK) Study
Acronym: Keifer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Therapeutic Area Head, Bayer Consumer Care Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 13080
Record Dates: First submitted 2008-06-05; First posted 2008-06-06 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-05

CONDITIONS: Bioavailability
Keywords: Naproxen Sodium
MeSH Terms: interventions — Naproxen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Other)
  Interventions: Drug: Naproxen sodium
- Arm 2 (Other)
  Interventions: Drug: Naproxen sodium

INTERVENTIONS:
Drug: Naproxen sodium — Administered under fasting condition
  Arms: Arm 1
Drug: Naproxen sodium — Administered under fed condition
  Arms: Arm 2

SUMMARY:
The purpose of this study is to provide information on how well an extended release formulation (a medication that is released and absorbed over a longer period of time than a regular release formulation of the medication) of naproxen sodium is absorbed into the bloodstream after eating a high calorie breakfast and also after fasting (not eating for 14 hours).

ELIGIBILITY:
Inclusion Criteria:

* Healthy, ambulatory, male and female volunteers between 18 to 55 years of age with a Body Mass Index (BMI) of approximately 18 to 30 kg/m2, and a total body weight > 50 kg (110 lbs);
* Results of screening and clinical laboratory tests are within normal range or considered not clinically significant by the Principal Investigator and the Sponsor;
* Female subjects of childbearing potential must be using a medically acceptable form of birth control for at least 1 month prior to screening (3 months on oral contraceptives), e.g., oral or patch contraceptives, intrauterine device, NuvaRing®, Depo-Provera®, or double-barrier and have a negative pregnancy test at Screening and Day 0 of each dosing period. Female subjects of nonchildbearing potential must be amenorrheic for at least 2 years or had a hysterectomy and/or bilateral oophorectomy

Exclusion Criteria:

* History of hypersensitivity to aspirin (ASA), naproxen sodium, or acetaminophen, and similar pharmacological agents or components of the products;
* Females who are pregnant or lactating;
* Loss of blood in excess of 500 ml within 56 days of the first dose of trial treatment (e.g., donation, plasmapheresis or injury);
* History of gastrointestinal bleeding or perforation, related to previous NSAID therapy. Active, or history of recurrent peptic ulcer/hemorrhage (two or more distinct episodes of proven ulceration or bleeding);
* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic diseases or malignancies;
* Positive alcohol or drug test;
* Have taken any medications (except acceptable forms of birth control) within 10 days prior to dosing or throughout the study, unless in the opinion of the Investigator and the Sponsor, the medication will not interfere with the study procedures, data integrity, or compromise the safety of the subject;
* Have taken ASA, ASA-containing products, acetaminophen (acetyl-para-amino-phenol or APAP) or any other NSAID (OTC or prescription) 7 days prior to dosing or during the treatment period, other than study treatment;
* Smokers or currently consuming any type of tobacco product(s) including any smoking cessation nicotine-containing product (e.g., nicotine patch, nicotine gum);
* Have taken any vitamin or herbal supplement within 7 days prior to dosing or refuse to refrain from use during the study;
* Alcoholism or drug abuse within 2 years prior to the Screening Visit;
* Participation in any other trials involving investigational or marketed products within 30 days prior to the Screening Visit.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2008-01; Primary Completion 2008-02 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
PK parameters | Over 48 hours

SECONDARY OUTCOMES:
Assess the tolerability of the investigational product. | Over 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Little Rock, Arkansas, United States